CLINICAL TRIAL: NCT00839657
Title: A Randomized, Multi-Center, Double-Blind Clinical Trial to Evaluate the Use of Clinical Plus Genetic Information to Guide Warfarin Therapy Initiation and Improve Anticoagulation Control for Patients
Brief Title: Clarification of Optimal Anticoagulation Through Genetics
Acronym: COAG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 623; N01 HV88210; HHSN268200800003C
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2013-05

CONDITIONS: Stroke; Venous Thrombosis; Atrial Fibrillation; Atrial Flutter
Keywords: Embolism; Thrombosis
MeSH Terms: conditions — Stroke; Venous Thrombosis; Atrial Fibrillation; Atrial Flutter; Embolism; Thrombosis | interventions — Warfarin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Genotype-guided dosing algorithm for warfarin
  Interventions: Behavioral: Genotype-guided dosing algorithm for warfarin
- 2 (Active Comparator): Clinical-guided dosing algorithm for warfarin
  Interventions: Behavioral: Clinical-guided dosing algorithm for warfarin

INTERVENTIONS:
Behavioral: Genotype-guided dosing algorithm for warfarin — Initial dosing of warfarin for the first 3-4 days of treatment will be determined by an algorithm that uses clinical and genetic information. Following this initiation dose of warfarin, a second dose adjustment will be made after 3 and/or 4 doses of warfarin using a dose revision algorithm that incorporates the clinical and genetic information.
  Arms: 1
Behavioral: Clinical-guided dosing algorithm for warfarin — Initial dosing of warfarin for the first 3-4 days of treatment will be determined by an algorithm that uses clinical information. Following this initiation dose of warfarin, a second dose adjustment will be made after 3 and/or 4 doses of warfarin using a dose revision algorithm that incorporates the clinical information.
  Arms: 2

SUMMARY:
Individuals taking warfarin often need frequent dose changes as the international normalized ratio (INR) gets too high or too low which could result in a higher risk of thromboembolism, bleeding and early discontinuation of a highly useful therapy. This study will compare two approaches to warfarin dosing to examine the utility of using genetic information for warfarin dosing.

DETAILED DESCRIPTION:
The objective of the Clarification of Optimal Anticoagulation through Genetics (COAG) trial is to conduct a 1,022 participant, multicenter, double-blind, randomized trial comparing two approaches to guiding warfarin therapy initiation: 1) initiation of warfarin therapy based on algorithms using clinical information and an individual's genotype using genes known to influence warfarin response ("genotype-guided dosing"), and 2) initiation of warfarin therapy based on algorithms using only clinical information ("clinical-guided dosing"). The study hypothesis is that the use of genetic and clinical information for selecting the dose of warfarin during the initial dosing period will lead to improvement in stability of anticoagulation(AC) relative to a strategy that incorporates only clinical information (without genetics) for initial dosing. Each study arm will include a baseline dose initiation algorithm and a dose revision algorithm applied over the first 4 to 5 doses of warfarin therapy. By comparing the two strategies in this trial, the study will be able to determine if genetic information provides added benefit above and beyond what can be gleaned simply with clinical information. This study is a proof-of-concept efficacy trial. Efficacy is defined as a measure of whether, under optimal application, dosing algorithms will lead to improvement in care. The trial will thus answer the question: "can the use of clinical plus genetic information lead to an improvement in anticoagulation control above and beyond the use of only clinical information during the initiation of warfarin, when applied in a uniform and optimal manner to all patients?" Because efficacy has not yet been established for genotype-guided dosing of warfarin, it is important to first test whether this approach can, indeed, improve anticoagulation outcomes under controlled conditions.

ELIGIBILITY:
Inclusion Criteria:

* Willingness and ability to sign informed consent
* Able to be followed in outpatient AC clinic
* Expected duration of warfarin therapy of at least 1 month
* AC management for the patient will be performed in-hospital and as an outpatient by clinicians that will adhere to the study dosing algorithms and dose titration plans
* Target INR 2-3

Exclusion Criteria:

* Currently taking warfarin
* Prior warfarin therapy with known required stable dose
* Clinician opinion that warfarin dosing needs to be adjusted for reasons not accounted for by dosing algorithm
* Abnormal baseline INR (off warfarin) (e.g., due to liver disease, antiphospholipid antibody)
* Contraindication to warfarin treatment for at least 3 months
* Life expectancy of less than 1 year
* Pregnant women or child-bearing women not using medically approved method of birth control (requires negative pregnancy test to exclude pregnancy in child-bearing women)
* Inability to follow-up on a regular basis with anticoagulation practitioners participating in the trial
* Any factors likely to limit adherence to warfarin
* Cognitive or other causes of inability to provide informed consent or follow study procedures
* Participating in another trial that prohibits participation in the COAG trial or planned enrollment in such a trial within the first 6 months of warfarin therapy
* Estimated blood loss of more than 1,000 cc requiring blood transfusions within 48 hours prior to randomization
* Genotype (CYP2C9 or VKORC1) known to participant from prior testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1015 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Percentage of time participants spend within the therapeutic INR range (PTTR) | Measured during the first 4 weeks of therapy

SECONDARY OUTCOMES:
Occurrence of INR greater than 4 or serious clinical event | Measured during the first 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen E Kimmel, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (18):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - Tulane University Health Science Center, New Orleans, Louisiana
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai School of Medicine, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health Care, Salt Lake City, Utah
  - Marshfield Clinical Research Foundation, Marshfield, Wisconsin

REFERENCES:
- [Background] Joo J, Geller NL, French B, Kimmel SE, Rosenberg Y, Ellenberg JH. Prospective alpha allocation in the Clarification of Optimal Anticoagulation through Genetics (COAG) trial. Clin Trials. 2010 Oct;7(5):597-604. doi: 10.1177/1740774510381285. Epub 2010 Aug 6. PMID 20693186
- [Background] Kimmel SE, French B, Anderson JL, Gage BF, Johnson JA, Rosenberg YD, Geller NL, Kasner SE, Eby CS, Joo J, Caldwell MD, Goldhaber SZ, Hart RG, Cifelli D, Madigan R, Brensinger CM, Goldberg S, Califf RM, Ellenberg JH. Rationale and design of the Clarification of Optimal Anticoagulation through Genetics trial. Am Heart J. 2013 Sep;166(3):435-41. doi: 10.1016/j.ahj.2013.04.009. Epub 2013 Jul 12. PMID 24016491
- [Result] Kimmel SE, French B, Kasner SE, Johnson JA, Anderson JL, Gage BF, Rosenberg YD, Eby CS, Madigan RA, McBane RB, Abdel-Rahman SZ, Stevens SM, Yale S, Mohler ER 3rd, Fang MC, Shah V, Horenstein RB, Limdi NA, Muldowney JA 3rd, Gujral J, Delafontaine P, Desnick RJ, Ortel TL, Billett HH, Pendleton RC, Geller NL, Halperin JL, Goldhaber SZ, Caldwell MD, Califf RM, Ellenberg JH; COAG Investigators. A pharmacogenetic versus a clinical algorithm for warfarin dosing. N Engl J Med. 2013 Dec 12;369(24):2283-93. doi: 10.1056/NEJMoa1310669. Epub 2013 Nov 19. PMID 24251361
- [Derived] French B, Joo J, Geller NL, Kimmel SE, Rosenberg Y, Anderson JL, Gage BF, Johnson JA, Ellenberg JH; COAG (Clarification of Optimal Anticoagulation through Genetics) Investigators. Statistical design of personalized medicine interventions: the Clarification of Optimal Anticoagulation through Genetics (COAG) trial. Trials. 2010 Nov 17;11:108. doi: 10.1186/1745-6215-11-108. PMID 21083927
- Available data/document: Individual Participant Data Set: COAG — http://biolincc.nhlbi.nih.gov/studies/coag/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/coag/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/coag/
- Available data/document: Manual of Procedures — http://biolincc.nhlbi.nih.gov/studies/coag/